CLINICAL TRIAL: NCT02983422
Title: Effects of Aminophylline on Renal Function and Urine Volume Acute Kidney Injury Patient
Brief Title: Effects of Aminophylline on Renal Function and Urine Volume of AKI Patient
Status: Unknown | Phase: Early Phase 1 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Shanghai Jiao Tong University Affiliated Sixth People's Hospital (Other)
Responsible Party: Principal Investigator, Gao Yanding, Deputy chief physician, Shanghai Jiao Tong University Affiliated Sixth People's Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: SSH-ICU-017
Record Dates: First submitted 2016-11-26; First posted 2016-12-06 (Estimated); Last update posted 2016-12-06 (Estimated); Status verified 2016-12

CONDITIONS: Acute Kidney Injury
MeSH Terms: conditions — Acute Kidney Injury | interventions — Aminophylline; Furosemide; Saline Solution

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Group aminophylline (Active Comparator): To increase the dose of frusemide until 15mg/h with Syringe pumps. If the urine doesn't reach 1ml/kg/h,then combined with Aminophylline(loading dose of 5mg/kg，and maintenance dose of 0.5mg/kg)
  Interventions: Drug: aminophylline; Drug: frusemide
- Group frusemide (Placebo Comparator): Use frusemide with Syringe pumps,maximum dose to 15mg/h，with placebo bolus followed by IV infusions of normal saline (0.9%) every hour (matched by volume and appearance to the treatment group)
  Interventions: Drug: frusemide; Drug: normal saline

INTERVENTIONS:
Drug: aminophylline — To increase the dose of frusemide until 15mg/h with Syringe pumps. If the urine doesn't reach 1ml/kg/h,then combined with Aminophylline(loading dose of 5mg/kg，and maintenance dose of 0.5mg/kg)
  Arms: Group aminophylline
Drug: frusemide — Use frusemide with Syringe pumps,maximum dose to 15mg/h
Drug: normal saline — Placebo bolus followed by IV infusions of normal saline (0.9%) every hour (matched by volume and appearance to the treatment group)
  Arms: Group frusemide

SUMMARY:
This study evaluates the effects of aminophylline on serum creatinine and urine volume of AKI Patient.Half of participants will receive aminophylline and furosemide in combination,while the other half will receive only furosemide.

DETAILED DESCRIPTION:
Acute kidney injury (AKI) is a sudden perturbation of kidney function that is frequently associated with high morbidity and mortality rates . A diagnostic time limit of 48 hours was recently introduced to ensure early diagnosis, management and prevention of progression to irreversible renal function loss . Furthermore, early AKI biomarkers that can ensure prompt diagnosis have been identified. When these biomarkers become widely available to clinical practice, informed therapeutic interventions capable of aborting disease progression, morbidity and mortality multiplication can be applied . In the injured kidney, adenosine is released endogenously from the macula densa causing vasoconstriction of the renal afferent arterioles via the adenosine A1receptor as well as vasodilatation of the renal efferent arterioles via the adenosine A2 receptor; thereby reducing the renal blood flow and glomerular perfusion pressure leading to ischemic kidney injury . One measure that has been tried with the objective of achieving better AKI outcome is the use of aminophylline (an ethylenediamine coupled theophylline) . Aminophylline is converted to theophylline in the human body, which in turn vasodilates the renal afferent arterioles through competitive inhibition of adenosine on the adenosine A1 receptor.

Aminophylline and theophylline, methylxanthine nonselective adenosine receptor antagonists, have been effective in the management of AKI in certain clinical scenarios including heart failure, calcineurin inhibitor toxicity, and perinatal asphyxia. In the kidney, adenosine constricts the afferent arteriole and decreases glomerular blood flow; adenosine receptor blockade mitigates this vasoconstriction. Aminophylline also inhibits phosphodiesterase at higher concentrations, which leads to increased urine output.

Eligible subjects included all patients more than 18 years old with acute kidney injury in ICU. To ensure the safest oversight for the duration of the study drug infusion, the investigators only approached patients for consent if participants' ICU stay would likely be at least 72 hours . Patients were recruited in the preoperative clinic or in the inpatient ward/ICU; the nature of the consent process for this interventional drug trial necessitated that all procedures were elective or scheduled. Because aminophylline has been associated with tachycardia and seizures at high serum levels, and its metabolism may be affected by liver or thyroid dysfunction and sepsis, the investigators selected the following exclusion criteria: history of tachyarrhythmias, seizures, coagulopathy (international normalized ratio > 1.5 while not taking warfarin),or hypothyroidism. Study investigators or research nurses recruited participants; written, informed consent was signed by each patient or guardian.

The treatment group received aminophylline 5 mg/kg IV load over 30 minutes, followed by 0.5 mg/kg IV every hour, for 72 hours .The control group received placebo bolus followed by IV infusions of normal saline (0.9%) every hour (matched by volume and appearance to the treatment group), for 72 hours.

ELIGIBILITY:
Inclusion Criteria:

* Patients with acute injury (AKI) with no lack of circulating volume (central venous pressure >8cmH2O)

Exclusion Criteria:

* Patients with chronic kidney disease
* Patients with acute renal injury caused by insufficient circulating volume
* Patients who do not cooperate with the use of the drug therapy
* Patients who do not cooperate with the relevant examination

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2016-12; Primary Completion 2017-06 (Estimated); Study Completion 2017-07 (Estimated)

PRIMARY OUTCOMES:
serum creatinine | Change from serum creatinine at 2 weeks
urine volume | Change from urine volume at 2 weeks
Serum cystatin-C | Change from Serum cystatin-C at 2 weeks
Urine β_2-microglobulin | Change from Urine β_2-microglobulin at 2 weeks

SECONDARY OUTCOMES:
dose of norepinephrine | Change from dose of norepinephrine at 2 weeks
blood pressure | Change from baseline systolic blood pressure at 2 weeks
central venous pressure | Change from central venous pressure at 2 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Xuemin Wang, PhD, Study Director — Shanghai 6th People's Hospital

REFERENCES:
- [Background] Parker MR, Willatts SM. A pilot study to investigate the effects of an infusion of aminophylline on renal function following major abdominal surgery. Anaesthesia. 2001 Jul;56(7):670-5. doi: 10.1046/j.1365-2044.2001.01374.x. PMID 11437769
- [Background] Lynch BA, Gal P, Ransom JL, Carlos RQ, Dimaguila MA, Smith MS, Wimmer JE Jr, Imm MD. Low-dose aminophylline for the treatment of neonatal non-oliguric renal failure-case series and review of the literature. J Pediatr Pharmacol Ther. 2008 Apr;13(2):80-7. doi: 10.5863/1551-6776-13.2.80. PMID 23055869
- [Background] Yang GZ, Xue FS, Liu GP, Sun C. Use of Aminophylline to Prevent Acute Kidney Injury After Pediatric Cardiac Surgery. Pediatr Crit Care Med. 2016 Aug;17(8):814. doi: 10.1097/PCC.0000000000000838. No abstract available. PMID 27500627
- [Background] Chen HH, Anstrom KJ, Givertz MM, Stevenson LW, Semigran MJ, Goldsmith SR, Bart BA, Bull DA, Stehlik J, LeWinter MM, Konstam MA, Huggins GS, Rouleau JL, O'Meara E, Tang WH, Starling RC, Butler J, Deswal A, Felker GM, O'Connor CM, Bonita RE, Margulies KB, Cappola TP, Ofili EO, Mann DL, Davila-Roman VG, McNulty SE, Borlaug BA, Velazquez EJ, Lee KL, Shah MR, Hernandez AF, Braunwald E, Redfield MM; NHLBI Heart Failure Clinical Research Network. Low-dose dopamine or low-dose nesiritide in acute heart failure with renal dysfunction: the ROSE acute heart failure randomized trial. JAMA. 2013 Dec 18;310(23):2533-43. doi: 10.1001/jama.2013.282190. PMID 24247300